CLINICAL TRIAL: NCT06300866
Title: The Clinical Investigation of Stannous Fluoride Containing Toothpaste Compared to Colgate Cavity Protection Toothpaste in Reducing Plaque and Gingivitis - a Six-month Study in California
Brief Title: Gingivitis Reduction After Use of 0.45% Stannous Fluoride Toothpaste
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRO-2020-04-PGN-LLU-YPZ
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Gingivitis; Plaque, Dental
Keywords: Loe and Silness Gingival Index; Quigley and Hein Plaque Index
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Experimental): toothpaste brushing 2x daily morning & evening for 2 minutes
  Interventions: Drug: Test; Drug: Control
- Group II (Active Comparator): toothpaste brushing 2x daily morning & evening for 2 minutes
  Interventions: Drug: Test; Drug: Control

INTERVENTIONS:
Drug: Test — test toothpaste containing 0.45% stannous fluoride
Drug: Control — toothpaste containing 0.76% sodium monofluorophosphate

SUMMARY:
The 6-month clinical study was designed to investigate clinical efficacy on plaque and gingivitis for the stannous fluoride containing toothpaste (SNAP) compared to Colgate Cavity Protection Toothpaste after 3 and 6 months of product use.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must meet all of the following criteria
* Subjects, ages 18-70, inclusive
* Availability for the six-month duration of the clinical research study
* Good general health
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe-Silness Gingival Index
* Initial plaque index of at least 1.5 as determined by the use of the Quigley-Hein Plaque Index
* Signed Informed Consent Form

Exclusion Criteria:

* Presence of orthodontic appliances
* Presence of partial removable dentures
* Tumor(s) of the soft or hard tissues of the oral cavity
* Moderate and/or advanced periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study
* Five or more carious lesions requiring immediate restorative treatment
* Antibiotic use any time during the one-month period prior to entry into the study -Participation in any other clinical study or test panel within the one month prior to entry into the study
* Dental prophylaxis during the past two weeks prior to baseline examinations
* History of allergies to oral care/personal care consumer products or their ingredients -On any prescription medicines that might interfere with the study outcome
* An existing medical condition that prohibits eating and/or drinking for periods up to 4 hours
* History of alcohol and/or drug abuse
* Self-reported pregnancy and/or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Whole-Mouth Gingivitis Measurement | baseline, 3 months and 6 months
  difference of reduction in gingival index
Whole-Mouth Dental Plaque Measurement | baseline, 3 months and 6 months
  difference of reduction in plaque index

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, DDS MSD PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No